CLINICAL TRIAL: NCT04713553
Title: A PHASE 3, RANDOMIZED, OBSERVER-BLIND STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF MULTIPLE PRODUCTION LOTS AND DOSE LEVELS OF THE VACCINE CANDIDATE BNT162b2 AGAINST COVID-19 IN HEALTHY PARTICIPANTS 12 THROUGH 50 YEARS OF AGE AND THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF BNT162b2 RNA-BASED COVID-19 VACCINE CANDIDATES AS A BOOSTER DOSE IN HEALTHY PARTICIPANTS 18 THROUGH 50 YEARS OF AGE
Brief Title: A Phase 3 Study to Evaluate the Safety, Tolerability, and Immunogenicity of Multiple Production Lots and Dose Levels of BNT162b2 RNA-Based COVID-19 Vaccines Against COVID-19 in Healthy Participants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: C4591017
Record Dates: First submitted 2021-01-15; First posted 2021-01-19 (Actual); Results first posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-11

CONDITIONS: SARS-CoV-2 Infection; COVID-19
Keywords: COVID-19; Coronavirus; Vaccine; SARS-CoV-2; RNA Vaccine; BNT162b2; BNT162B2.1.B.351
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — BNT162 Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Arm 1 (Experimental): 30-microgram dose of US manufactured drug substance (Lot 1)
  Interventions: Biological: BNT162b2
- Arm 2 (Experimental): 30-microgram dose of US manufactured drug substance (Lot 2)
  Interventions: Biological: BNT162b2
- Arm 3 (Experimental): 30-microgram dose of US manufactured drug substance (Lot 3)
  Interventions: Biological: BNT162b2
- Arm 4 (Experimental): 30-microgram dose of EU manufactured drug substance (Lot 4)
  Interventions: Biological: BNT162b2
- Arm 5 (Experimental): 20-microgram dose of US manufactured drug substance (corresponding to Arm 1, 2 or 3 lot)
  Interventions: Biological: BNT162b2
- Booster 1: BNT162b2 (Experimental): 30-microgram dose
  Interventions: Biological: BNT162b2
- Booster 2: BNT162b2.B.1.351 (Experimental): 30-microgram dose
  Interventions: Biological: BNT162b2.B.1.351

INTERVENTIONS:
Biological: BNT162b2 — Intramuscular injection
  Arms: Arm 1; Arm 2; Arm 3; Arm 4; Arm 5; Booster 1: BNT162b2
Biological: BNT162b2.B.1.351 — Intramuscular injection
  Arms: Booster 2: BNT162b2.B.1.351

SUMMARY:
This is a Phase 3, randomized, observer-blind study in healthy individuals.

The primary study will evaluate the safety, tolerability, and immunogenicity of the SARS-CoV-2 RNA vaccine candidate (BNT162b2):

* As a 30-microgram dose, administered from 1 of 4 manufacturing lots (batches)
* As a 20-microgram dose, administered from 1 of the manufacturing lots
* As a 2-dose (separated by 21 days) schedule
* In people 12 through 50 years of age

The booster study will evaluate the safety, tolerability, and immunogenicity of 2 SARS-CoV-2 RNA vaccine candidates (BNT162b2 and BNT162b2.B.1.351):

* Each as a 30-microgram dose
* Each as a 1-dose booster vaccine, administered approximately 3 months after Dose 2
* In people 18 through 50 years of age

ELIGIBILITY:
Inclusion Criteria:

* Primary study: Male or female participants between the ages of 12 and 50 years, inclusive, at randomization.
* Booster study: Male or female participants between the ages of 18 and 50 years, inclusive, at rerandomization.
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
* Healthy participants who are determined by medical history, physical examination (if required), and clinical judgment of the investigator to be eligible for inclusion in the study.
* Capable of giving personal signed informed consent/have parent(s)/legal guardian capable of giving signed informed consent.

Exclusion Criteria:

* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Known infection with HIV, HCV, or HBV.
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention.
* Previous clinical (based on COVID-19 symptoms/signs alone, if a SARS-CoV-2 NAAT result was not available) or microbiological (based on COVID-19 symptoms/signs and a positive SARS-CoV-2 NAAT result) diagnosis of COVID 19.

  . Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
* Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
* Women who are pregnant or breastfeeding.
* Primary study: Previous vaccination with any coronavirus vaccine.
* Booster study: Previous vaccination with any coronavirus vaccine outside of this study.
* Receipt of medications intended to prevent COVID-19.
* Individuals who receive treatment with radiotherapy or immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids, eg, for cancer or an autoimmune disease, or planned receipt throughout the study.
* Receipt of blood/plasma products or immunoglobulin, from 60 days before study intervention administration or planned receipt throughout the study.
* Participation in other studies involving study intervention within 28 days prior to study entry and/or during study participation.
* Previous participation in other studies involving study intervention containing lipid nanoparticles.
* Investigator site staff or Pfizer/BioNTech employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

Additional Exclusion Criteria for the Booster study:

* Current febrile illness (body temperature ≥100.4°F [≥38.0°C]) or other acute illness within 48 hours before study intervention administration.
* Receipt of any seasonal or pandemic influenza vaccine within 14 days, or any other nonstudy vaccine within 28 days, before or after study intervention administration.
* Receipt of short-term (<14 days) systemic corticosteroids. Inhaled/nebulized, intra-articular, intrabursal, or topical (skin or eyes) corticosteroids are permitted.

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1574 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-07-22 (Actual); Study Completion 2021-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (16):
- United States (16):
  - Kaiser Permanente Oakland, Oakland, California
  - Clinical Research Consulting, Milford, Connecticut
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - Research Centers of America, Hollywood, Florida
  - Clinical Neuroscience Solutions, Orlando, Florida
  - Clinical Research Atlanta, Stockbridge, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Solaris Clinical Research, Meridian, Idaho
  - Kentucky Pediatric/Adult Research, Bardstown, Kentucky
  - Amici Clinical Research LLC, Raritan, New Jersey
  - Accellacare - Wilmington, Wilmington, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Texas Center for Drug Development, Inc., Houston, Texas
  - Clinical Trials of Texas, LLC, San Antonio, Texas
  - Martin Diagnostic Clinic, Tomball, Texas
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4591017

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in two parts: primary study and booster study.
Pre-assignment Details: Total number of participants enrolled in study and assigned to study intervention were 1574, however, only 1573 participants received study intervention.
Groups:
- BNT162b2 30 mcg: US Lot 1: Participants were randomized in primary study to receive 30 microgram (mcg) intramuscular dose of BNT162b2 (US Lot 1) vaccine as 2-dose schedule separated by 21 days. Participants were followed up for safety for up to 28-35 days after second dose of vaccine, for a maximum of 2 months.
- BNT162b2 30 mcg: US Lot 2: Participants were randomized in primary study to receive 30 mcg intramuscular dose of BNT162b2 (US Lot 2) vaccine as 2-dose schedule separated by 21 days. Participants were followed up for safety for up to 28-35 days after second dose of vaccine, for a maximum of 2 months.
- BNT162b2 30 mcg: US Lot 3: Participants were randomized in primary study to receive 30 mcg intramuscular dose of BNT162b2 (US Lot 3) vaccine as 2-dose schedule separated by 21 days. Participants were followed up for safety for up to 28-35 days after second dose of vaccine, for a maximum of 2 months.
- BNT162b2 30 mcg: EU Lot: Participants were randomized in primary study to receive 30 mcg intramuscular dose of BNT162b2 (EU Lot) vaccine as 2-dose schedule separated by 21 days. Participants were followed up for safety for up to 28-35 days after second dose of vaccine, for a maximum of 2 months.
- BNT162b2 20 mcg: US Lot 1: Participants were randomized in primary study to receive 20 mcg intramuscular dose of BNT162b2 vaccine as 2-dose schedule separated by 21 days. Participants were followed up for safety for up to 28-35 days after second dose of vaccine, for a maximum of 2 months.
- BNT162b2 30 mcg: Booster Dose: Participants who received 2 doses of 30 mcg BNT162b2 vaccine in primary study from US Lot 1 were randomized to booster study to receive a single 30 mcg intramuscular dose of BNT162b2 vaccine at 3 months after second dose in the primary study. Participants were followed up for safety for up to 28-35 days after vaccination.
- BNT162b2.B.1.351 30 mcg: Booster Dose: Participants who received 2 doses of 30 mcg BNT162b2 vaccine in primary study from US Lot 1, 2 or 3 were randomized to booster study to receive a single 30 mcg intramuscular dose of BNT162b2.B.1.351 vaccine at 3 months after second dose in the primary study. Participants were followed up for safety for up to 28-35 days after vaccination.
Period: Primary Study (2 Months)
Arm/Group | BNT162b2 30 mcg: US Lot 1 | BNT162b2 30 mcg: US Lot 2 | BNT162b2 30 mcg: US Lot 3 | BNT162b2 30 mcg: EU Lot | BNT162b2 20 mcg: US Lot 1 | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Started | 351 | 352 | 347 | 173 | 351 | 0 (No participants were enrolled in this arm during the primary study.) | 0 (No participants were enrolled in this arm during the primary study.)
Treated | 351 | 352 | 346 | 173 | 351 | 0 | 0
Completed | 347 | 346 | 344 | 171 | 349 | 0 | 0
Not Completed | 4 | 6 | 3 | 2 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by parent/guardian | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Other | 1 | 2 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 2 | 1 | 0 | 0 | 0
Not completed — Inclusion criteria not met | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Booster Study (1 Month)
Arm/Group | BNT162b2 30 mcg: US Lot 1 | BNT162b2 30 mcg: US Lot 2 | BNT162b2 30 mcg: US Lot 3 | BNT162b2 30 mcg: EU Lot | BNT162b2 20 mcg: US Lot 1 | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Started | 0 | 0 | 0 | 0 | 0 | 31 | 31
Completed | 0 | 0 | 0 | 0 | 0 | 31 | 31
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population comprising of all randomized participants who received at least 1 dose of the study intervention were included.
Groups:
- BNT162b2 30 mcg: US Lot 1: Participants were randomized in primary study to receive 30 mcg intramuscular dose of BNT162b2 (US Lot 1) vaccine as 2-dose schedule separated by 21 days. Participants were followed up for safety for up to 28-35 days after second dose of vaccine, for a maximum of 2 months.
- Total: Total of all reporting groups
Arm/Group | BNT162b2 30 mcg: US Lot 1 | BNT162b2 30 mcg: US Lot 2 | BNT162b2 30 mcg: US Lot 3 | BNT162b2 30 mcg: EU Lot | BNT162b2 20 mcg: US Lot 1 | Total
Number analyzed (Participants) | 351 | 352 | 346 | 173 | 351 | 1573
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.0 (11.66) | 27.8 (11.76) | 27.5 (11.54) | 27.7 (11.40) | 27.5 (11.71) | 27.7 (11.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 177 | 176 | 159 | 83 | 163 | 758
  Male | 174 | 176 | 187 | 90 | 188 | 815
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 44 | 32 | 55 | 22 | 42 | 195
  Not Hispanic or Latino | 306 | 319 | 291 | 151 | 309 | 1376
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 0 | 3 | 5
  Asian | 36 | 48 | 40 | 24 | 44 | 192
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 1 | 0 | 2 | 5
  Black or African American | 21 | 16 | 15 | 2 | 14 | 68
  White | 286 | 280 | 283 | 142 | 283 | 1274
  More than one race | 6 | 5 | 5 | 4 | 5 | 25
  Unknown or Not Reported | 1 | 1 | 1 | 1 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Ratios (GMRs) of Full-Length S-Binding Immunoglobulin G (IgG) Concentrations Between Individual US Lots 1, 2, and 3 at 1 Month After Dose 2: Primary Study
Description: Geometric mean concentration of full-length S-binding IgG level for individual US lots (US lots 1, 2, and 3) was determined and reported in the descriptive section. Assay results below the lower limit of quantitation (LLOQ) were set to 0.5*LLOQ. GMRs were reported in the statistical analysis section and was calculated as ratio of Geometric Mean Concentrations (GMCs) of individual US Lots BNT162b2 30 mcg: US Lot 1, BNT162b2 30 mcg: US Lot 2 and BNT162b2 30 mcg: US Lot 3.
Time Frame: 1 Month after Dose 2
Population: Evaluable immunogenicity population: Participants who received 2 doses of vaccine in primary study, with Dose 2 received within predefined window, had at least 1 valid immunogenicity result from blood sample collected within an appropriate window at 1 month after Dose 2, were negative for both SARS-CoV-2 test (RT-PCR and N-blinding antibody) during study and had no other protocol deviations determined by clinician. Here, "N"= participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Unit per milliliter
Arm/Group | BNT162b2 30 mcg: US Lot 1 | BNT162b2 30 mcg: US Lot 2 | BNT162b2 30 mcg: US Lot 3
Number analyzed (Participants) | 324 | 311 | 310
Unit per milliliter | 6299.5 (5835.4) [5835.4 to 6800.5] | 6231.9 (5763.7) [5763.7 to 6738.2] | 6774.8 (6264.9) [6264.9 to 7326.1]
Statistical Analysis 1: Comparison: BNT162b2 30 mcg: US Lot 1 vs BNT162b2 30 mcg: US Lot 2; Test type: Equivalence — Equivalence was to be achieved if the 2-sided 95% confidence interval (CI) for GMR falls within the interval (0.67, 1.5); Geometric mean ratio = 1.01, 95% CI 2-sided [0.91 to 1.13] — GMRs and corresponding 2-sided 95% CIs were calculated by exponentiating difference in LS means and corresponding CIs based on analysis of logarithmically transformed assay results using a linear regression model with terms of age and vaccine group
Statistical Analysis 2: Comparison: BNT162b2 30 mcg: US Lot 1 vs BNT162b2 30 mcg: US Lot 3; Test type: Equivalence — Equivalence was to be achieved if the 2-sided 95% CI for GMR falls within the interval (0.67, 1.5); Geometric mean ratio = 0.93, 95% CI 2-sided [0.83 to 1.04] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: BNT162b2 30 mcg: US Lot 2 vs BNT162b2 30 mcg: US Lot 3; Test type: Equivalence — Equivalence was to be achieved if the 2-sided 95% CI for GMR falls within the interval (0.67, 1.5); Geometric mean ratio = 0.92, 95% CI 2-sided [0.82 to 1.03] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Geometric Mean Ratios (GMRs) of Full-Length S-Binding IgG Concentrations Between EU Lot and Pooled US Lots at 1 Month After Dose 2: Primary Study
Description: Geometric mean concentration of full-length S-binding IgG level for EU lot and pooled US lots (BNT162b2 30 mcg: US Lot 1, BNT162b2 30 mcg: US Lot 2 and BNT162b2 30 mcg: US Lot 3 reporting arm) were determined and reported in the descriptive section. Assay results below the LLOQ were set to 0.5*LLOQ. GMRs were reported in the statistical analysis section and was calculated as ratios of GMCs of BNT162b2 30 mcg: EU Lot and pooled US Lots (BNT162b2 30 mcg: US Lot 1, BNT162b2 30 mcg: US Lot 2 and BNT162b2 30 mcg: US Lot 3 reporting arm).
Time Frame: 1 Month after Dose 2
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Unit per milliliter
Groups:
- Pooled US Lots: Participants randomized in primary study to receive 30 mcg intramuscular dose of BNT162b2 (US Lot 1 + US Lot 2 + US Lot 3) vaccine as 2-dose schedule separated by 21 days. Participants were followed up for safety for up to 28-35 days after second dose of vaccine, for a maximum of 2 months.
Arm/Group | BNT162b2 30 mcg: EU Lot | Pooled US Lots
Number analyzed (Participants) | 160 | 945
Unit per milliliter | 6098.6 [5474.7 to 6793.7] | 6428.8 [6149.5 to 6720.7]
Statistical Analysis 1: Comparison: BNT162b2 30 mcg: EU Lot vs Pooled US Lots; Test type: Equivalence — Equivalence was to be achieved if the 2-sided 95% CI for GMR falls within the interval (0.67, 1.5); Geometric mean ratio = 0.95, 95% CI 2-sided [0.84 to 1.07] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Geometric Mean Ratios (GMRs) of SARS-CoV-2 Neutralizing Titers Between 20-microgram Dose and 30-microgram Dose at 1 Month After Dose 2: Primary Study
Description: Geometric mean titer for SARS-CoV-2 neutralizing titers for 20 mcg dose and 30 mcg dose of US Lot 1 was determined and reported in the descriptive section. GMTs and 2-sided 95% CIs were calculated by exponentiating the least square (LS) mean of the titers and corresponding CIs based on linear regression model. Assay results below the LLOQ were set to 0.5*LLOQ. GMRs were reported in the statistical analysis section and were calculated as the ratio of geometric mean titer of the 20-mcg dose (US Lot 1) to the geometric mean titer of the 30 mcg dose (US Lot 1).
Time Frame: 1 Month after Dose 2
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | BNT162b2 30 mcg: US Lot 1 | BNT162b2 20 mcg: US Lot 1
Number analyzed (Participants) | 318 | 324
Titer | 906.3 [847.8 to 968.9] | 976.6 [914.1 to 1043.4]
Statistical Analysis 1: Comparison: BNT162b2 30 mcg: US Lot 1 vs BNT162b2 20 mcg: US Lot 1; Test type: Non-Inferiority — Noninferiority of the 20 mcg dose to the corresponding 30 mcg dose was said to be achieved if the lower limit of the 2-sided 95% CI for the GMR is >0.67; Geometric Mean Ratio = 0.93, 95% CI 2-sided [0.84 to 1.02] — GMRs were calculated by exponentiating the difference in LS means and corresponding CIs based on analysis of logarithmically transformed assay results using a linear regression model with terms of age and vaccine group

4. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Dose 1: Primary Study
Description: Local reactions were collected by the participant using an electronic diary. Local reactions included redness, swelling, and pain at injection site after Dose 1. Redness, swelling, and pain at injection site after Dose 1 were reported.
Time Frame: Within 7 days after Dose 1
Population: Safety population included all randomized participants who received at least 1 dose of the study intervention. Here, "Overall Number of Participants Analyzed"= participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BNT162b2 30 mcg: US Lot 1 | BNT162b2 30 mcg: US Lot 2 | BNT162b2 30 mcg: US Lot 3 | Pooled US Lots | BNT162b2 30 mcg: EU Lot | BNT162b2 20 mcg: US Lot 1
Number analyzed (Participants) | 351 | 352 | 345 | 1048 | 173 | 351
Percentage of participants
  Redness | 1.1 [0.3 to 2.9] | 2.0 [0.8 to 4.1] | 2.9 [1.4 to 5.3] | 2.0 [1.2 to 3.0] | 2.3 [0.6 to 5.8] | 2.0 [0.8 to 4.1]
  Swelling | 2.0 [0.8 to 4.1] | 3.7 [2.0 to 6.2] | 3.8 [2.0 to 6.4] | 3.1 [2.2 to 4.4] | 2.9 [0.9 to 6.6] | 3.4 [1.8 to 5.9]
  Pain at Injection Site | 82.9 [78.6 to 86.7] | 79.3 [74.6 to 83.4] | 84.6 [80.4 to 88.3] | 82.3 [79.8 to 84.5] | 86.1 [80.1 to 90.9] | 78.1 [73.4 to 82.3]

5. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Dose 2: Primary Study
Description: Local reactions were collected by the participant using an electronic diary. Local reactions included redness, swelling, and pain at injection site after Dose 2. Redness, swelling, and pain at injection site after Dose 2 were reported.
Time Frame: Within 7 days after Dose 2
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BNT162b2 30 mcg: US Lot 1 | BNT162b2 30 mcg: US Lot 2 | BNT162b2 30 mcg: US Lot 3 | Pooled US Lots | BNT162b2 30 mcg: EU Lot | BNT162b2 20 mcg: US Lot 1
Number analyzed (Participants) | 349 | 350 | 343 | 1042 | 172 | 348
Percentage of participants
  Redness | 3.7 [2.0 to 6.3] | 4.0 [2.2 to 6.6] | 4.4 [2.5 to 7.1] | 4.0 [2.9 to 5.4] | 2.9 [1.0 to 6.7] | 3.2 [1.6 to 5.6]
  Swelling | 4.9 [2.9 to 7.7] | 6.0 [3.8 to 9.0] | 4.7 [2.7 to 7.5] | 5.2 [3.9 to 6.7] | 3.5 [1.3 to 7.4] | 3.7 [2.0 to 6.3]
  Pain at Injection Site | 80.2 [75.7 to 84.3] | 77.7 [73.0 to 82.0] | 83.1 [78.7 to 86.9] | 80.3 [77.8 to 82.7] | 77.3 [70.3 to 83.4] | 79.6 [75.0 to 83.7]

6. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Any Dose: Primary Study
Description: Local reactions were collected by the participant using an electronic diary. Local reactions included redness, swelling, and pain at injection site after each vaccination. Redness, swelling, and pain at injection site after any dose were reported.
Time Frame: Within 7 days after any dose
Population: Safety population included all randomized participants who received at least 1 dose of the study intervention. 1 participant randomized to US Lot 1 was administered US Lot 1 for Dose 1 and US Lot 3 for Dose 2, therefore, the participant was included in both reporting groups (US Lot 1 and US Lot 3).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BNT162b2 30 mcg: US Lot 1 | BNT162b2 30 mcg: US Lot 2 | BNT162b2 30 mcg: US Lot 3 | Pooled US Lots | BNT162b2 30 mcg: EU Lot | BNT162b2 20 mcg: US Lot 1
Number analyzed (Participants) | 351 | 352 | 347 | 1049 | 173 | 351
Percentage of participants
  Redness | 4.6 [2.6 to 7.3] | 5.4 [3.3 to 8.3] | 6.6 [4.2 to 9.8] | 5.5 [4.2 to 7.1] | 4.6 [2.0 to 8.9] | 4.6 [2.6 to 7.3]
  Swelling | 6.0 [3.7 to 9.0] | 8.8 [6.1 to 12.3] | 7.2 [4.7 to 10.5] | 7.3 [5.8 to 9.1] | 4.6 [2.0 to 8.9] | 6.3 [4.0 to 9.3]
  Pain at Injection Site | 90.9 [87.4 to 93.7] | 85.8 [81.7 to 89.3] | 91.1 [87.6 to 93.8] | 89.2 [87.2 to 91.0] | 91.3 [86.1 to 95.1] | 89.5 [85.8 to 92.5]

7. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Dose 3: Booster Study
Description: Local reactions were collected by the participant using an electronic diary. Local reactions included redness, swelling, and pain at injection site after Dose 3. Redness, swelling, and pain at injection site after Dose 3 were reported.
Time Frame: Within 7 days after Dose 3
Population: Safety population included all randomized participants who received dose 3 of the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Number analyzed (Participants) | 31 | 31
Percentage of participants
  Redness | 9.7 (2.0) [2.0 to 25.8] | 3.2 (0.1) [0.1 to 16.7]
  Swelling | 6.5 (0.8) [0.8 to 21.4] | 6.5 (0.8) [0.8 to 21.4]
  Pain at Injection site | 90.3 (74.2) [74.2 to 98.0] | 93.5 (78.6) [78.6 to 99.2]

8. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Dose 1: Primary Study
Description: Systemic events were reported using an electronic diary. Fever was defined as temperature >=38.0 degree Celsius (C) and categorized as >=38.0 to 38.4 C; >38.4 to 38.9 C; >38.9 to 40.0 C; >40.0 C. Systemic events including fever, fatigue, headache, chills, new or worsened muscle pain, new or worsened joint pain, vomiting, diarrhea, and use of antipyretic/analgesic medication after Dose 1 were reported.
Time Frame: Within 7 days after Dose 1
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BNT162b2 30 mcg: US Lot 1 | BNT162b2 30 mcg: US Lot 2 | BNT162b2 30 mcg: US Lot 3 | Pooled US Lots | BNT162b2 30 mcg: EU Lot | BNT162b2 20 mcg: US Lot 1
Number analyzed (Participants) | 351 | 352 | 345 | 1048 | 173 | 351
Percentage of participants
  Fever >=38.0 C | 0.3 [0.0 to 1.6] | 0 [0.0 to 1.0] | 2.0 [0.8 to 4.1] | 0.8 [0.3 to 1.5] | 1.2 [0.1 to 4.1] | 0 [0.0 to 1.0]
  Fever >=38.0 C to 38.4 C | 0.3 [0.0 to 1.6] | 0 [0.0 to 1.0] | 1.2 [0.3 to 2.9] | 0.5 [0.2 to 1.1] | 0.6 [0.0 to 3.2] | 0 [0.0 to 1.0]
  Fever >38.4 C to 38.9 C | 0 [0.0 to 1.0] | 0 [0.0 to 1.0] | 0.6 [0.1 to 2.1] | 0.2 [0.0 to 0.7] | 0.6 [0.0 to 3.2] | 0 [0.0 to 1.0]
  Fever >38.9 C to 40.0 C | 0 [0.0 to 1.0] | 0 [0.0 to 1.0] | 0.3 [0.0 to 1.6] | 0.1 [0.0 to 0.5] | 0 [0.0 to 2.1] | 0 [0.0 to 1.0]
  Fever >40.0 C | 0 [0.0 to 1.0] | 0 [0.0 to 1.0] | 1 [0.0 to 1.1] | 0 [0.0 to 0.4] | 0 [0.0 to 2.1] | 0 [0.0 to 1.0]
  Fatigue | 53.3 [47.9 to 58.6] | 45.5 [40.2 to 50.8] | 50.7 [45.3 to 56.1] | 49.8 [46.7 to 52.9] | 49.1 [41.5 to 56.8] | 49.0 [43.7 to 54.4]
  Headache | 36.2 [31.1 to 41.5] | 32.7 [27.8 to 37.8] | 33.3 [28.4 to 38.6] | 34.1 [31.2 to 37.0] | 38.7 [31.4 to 46.4] | 35.6 [30.6 to 40.9]
  Chills | 8.5 [5.8 to 12.0] | 7.7 [5.1 to 11.0] | 10.1 [7.2 to 13.8] | 8.8 [7.1 to 10.7] | 8.1 [4.5 to 13.2] | 6.8 [4.4 to 10.0]
  Vomiting | 0.6 [0.1 to 2.0] | 0.6 [0.1 to 2.0] | 1.2 [0.3 to 2.9] | 0.8 [0.3 to 1.5] | 0.6 [0.0 to 3.2] | 0.9 [0.2 to 2.5]
  Diarrhea | 9.7 [6.8 to 13.3] | 8.0 [5.4 to 11.3] | 7.8 [5.2 to 11.2] | 8.5 [6.9 to 10.3] | 9.2 [5.4 to 14.6] | 10.0 [7.0 to 13.6]
  New/worsened muscle pain | 14.5 [11.0 to 18.7] | 13.1 [9.7 to 17.0] | 16.5 [12.8 to 20.9] | 14.7 [12.6 to 17.0] | 17.3 [12.0 to 23.8] | 16.2 [12.5 to 20.5]
  New/worsened joint pain | 6.8 [4.4 to 10.0] | 6.5 [4.2 to 9.6] | 7.0 [4.5 to 10.2] | 6.8 [5.3 to 8.5] | 7.5 [4.1 to 12.5] | 6.6 [4.2 to 9.7]
  Use of antipyretic/analgesic medication | 16.8 [13.0 to 21.1] | 14.5 [11.0 to 18.6] | 18.8 [14.9 to 23.4] | 16.7 [14.5 to 19.1] | 22.0 [16.0 to 28.9] | 18.2 [14.3 to 22.7]

9. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Dose 2: Primary Study
Description: Systemic events were reported using an electronic diary. Fever was defined as temperature >=38.0 C and categorized as >=38.0 to 38.4 C; >38.4 to 38.9 C; >38.9 to 40.0 C; >40.0 C. Systemic events including fever, fatigue, headache, chills, new or worsened muscle pain, new or worsened joint pain, vomiting, diarrhea, and use of antipyretic/analgesic medication after Dose 2 were reported.
Time Frame: Within 7 days after Dose 2
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BNT162b2 30 mcg: US Lot 1 | BNT162b2 30 mcg: US Lot 2 | BNT162b2 30 mcg: US Lot 3 | Pooled US Lots | BNT162b2 30 mcg: EU Lot | BNT162b2 20 mcg: US Lot 1
Number analyzed (Participants) | 349 | 350 | 343 | 1042 | 172 | 348
Percentage of participants
  Fever >=38.0 C | 7.2 [4.7 to 10.4] | 6.3 [4.0 to 9.4] | 6.7 [4.3 to 9.9] | 6.7 [5.3 to 8.4] | 8.7 [5.0 to 14.0] | 5.7 [3.5 to 8.7]
  Fever >=38.0 C to 38.4 C | 4.6 [2.6 to 7.3] | 3.4 [1.8 to 5.9] | 3.2 [1.6 to 5.7] | 3.7 [2.7 to 5.1] | 6.4 [3.2 to 11.2] | 4.3 [2.4 to 7.0]
  Fever >38.4 C to 38.9 C | 2.0 [0.8 to 4.1] | 2.0 [0.8 to 4.1] | 2.3 [1.0 to 4.5] | 2.1 [1.3 to 3.2] | 1.2 [0.1 to 4.1] | 1.4 [0.5 to 3.3]
  Fever >38.9 C to 40.0 C | 0.6 [0.1 to 2.1] | 0.9 [0.2 to 2.5] | 0.9 [0.2 to 2.5] | 0.8 [0.3 to 1.5] | 1.2 [0.1 to 4.1] | 0 [0.0 to 1.1]
  Fever >40.0 C | 0 [0.0 to 1.1] | 0 [0.0 to 1.0] | 0.3 [0.0 to 1.6] | 0.1 [0.0 to 0.5] | 0 [0.0 to 2.1] | 0 [0.0 to 2.1]
  Fatigue | 69.9 [64.8 to 74.7] | 66.6 [61.4 to 71.5] | 71.4 [66.3 to 76.2] | 69.3 [66.4 to 72.1] | 69.8 [62.3 to 76.5] | 66.7 [61.4 to 71.6]
  Headache | 57.0 [51.6 to 62.3] | 56.6 [51.2 to 61.8] | 56.9 [51.4 to 62.2] | 56.8 [53.7 to 59.8] | 56.4 [48.6 to 63.9] | 50.6 [45.2 to 55.9]
  Chills | 28.1 [23.4 to 33.1] | 31.1 [26.3 to 36.3] | 33.8 [28.8 to 39.1] | 31.0 [28.2 to 33.9] | 28.5 [21.9 to 35.9] | 23.6 [19.2 to 28.4]
  Vomiting | 2.3 [1.0 to 4.5] | 1.4 [0.5 to 3.3] | 2.3 [1.0 to 4.5] | 2.0 [1.3 to 3.1] | 1.7 [0.4 to 5.0] | 1.4 [0.5 to 3.3]
  Diarrhea | 8.3 [5.6 to 11.7] | 9.1 [6.3 to 12.7] | 7.9 [5.3 to 11.2] | 8.4 [6.8 to 10.3] | 9.3 [5.4 to 14.7] | 6.9 [4.5 to 10.1]
  New/worsened muscle pain | 32.7 [27.8 to 37.9] | 38.6 [33.4 to 43.9] | 35.6 [30.5 to 40.9] | 35.6 [32.7 to 38.6] | 36.0 [28.9 to 43.7] | 35.6 [30.6 to 40.9]
  New/worsened joint pain | 19.2 [15.2 to 23.7] | 24.6 [20.2 to 29.4] | 19.2 [15.2 to 23.8] | 21.0 [18.6 to 23.6] | 19.2 [13.6 to 25.9] | 19.5 [15.5 to 24.1]
  Use of antipyretic/analgesic medication | 35.2 [30.2 to 40.5] | 41.1 [35.9 to 46.5] | 40.8 [35.6 to 46.2] | 39.1 [36.1 to 42.1] | 41.9 [34.4 to 49.6] | 37.9 [32.8 to 43.3]

10. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Any Dose: Primary Study
Description: Systemic events were reported using an electronic diary. Fever was defined as temperature >=38.0 C and categorized as >=38.0 to 38.4 C; >38.4 to 38.9 C; >38.9 to 40.0 C; >40.0 C. Systemic events including fever, fatigue, headache, chills, new or worsened muscle pain, new or worsened joint pain, vomiting, diarrhea, and use of antipyretic/analgesic medication after any dose were reported.
Time Frame: Within 7 days after any dose
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BNT162b2 30 mcg: US Lot 1 | BNT162b2 30 mcg: US Lot 2 | BNT162b2 30 mcg: US Lot 3 | Pooled US Lots | BNT162b2 30 mcg: EU Lot | BNT162b2 20 mcg: US Lot 1
Number analyzed (Participants) | 351 | 352 | 347 | 1049 | 173 | 351
Percentage of participants
  Fever >=38.0 C | 7.4 [4.9 to 10.7] | 6.3 [4.0 to 9.3] | 8.4 [5.7 to 11.8] | 7.3 [5.8 to 9.1] | 9.2 [5.4 to 14.6] | 5.7 [3.5 to 8.7]
  Fever >=38.0 C to 38.4 C | 4.8 [2.8 to 7.6] | 3.4 [1.8 to 5.9] | 4.0 [2.2 to 6.7] | 4.1 [3.0 to 5.5] | 6.4 [3.2 to 11.1] | 4.3 [2.4 to 7.0]
  Fever >38.4 C to 38.9 C | 2.0 [0.8 to 4.1] | 2.0 [0.8 to 4.1] | 2.9 [1.4 to 5.2] | 2.3 [1.5 to 3.4] | 1.7 [0.4 to 5.0] | 1.4 [0.5 to 3.3]
  Fever >38.9 C to 40.0 C | 0.6 [0.1 to 2.0] | 0.9 [0.2 to 2.5] | 1.2 [0.3 to 2.9] | 0.9 [0.4 to 1.6] | 1.2 [0.1 to 4.1] | 0 [0.0 to 1.0]
  Fever >40.0 C | 0 [0.0 to 1.0] | 0 [0.0 to 1.0] | 0.3 [0.0 to 1.6] | 0.1 [0.0 to 0.5] | 0 [0.0 to 2.1] | 0 [0.0 to 1.0]
  Fatigue | 78.6 [74.0 to 82.8] | 73.6 [68.6 to 78.1] | 81.0 [76.4 to 85.0] | 77.8 [75.1 to 80.3] | 76.9 [69.9 to 82.9] | 75.5 [70.7 to 79.9]
  Headache | 66.7 [61.5 to 71.6] | 65.1 [59.8 to 70.0] | 64.3 [59.0 to 69.3] | 65.4 [62.4 to 68.3] | 68.8 [61.3 to 75.6] | 63.8 [58.5 to 68.9]
  Chills | 32.8 [27.9 to 37.9] | 34.1 [29.1 to 39.3] | 37.2 [32.1 to 42.5] | 34.7 [31.8 to 37.7] | 32.4 [25.5 to 39.9] | 26.2 [21.7 to 31.1]
  Vomiting | 2.8 [1.4 to 5.2] | 2.0 [0.8 to 4.1] | 3.5 [1.8 to 6.0] | 2.8 [1.9 to 3.9] | 2.3 [0.6 to 5.8] | 2.3 [1.0 to 4.4]
  Diarrhea | 16.2 [12.5 to 20.5] | 14.2 [10.7 to 18.3] | 13.8 [10.4 to 17.9] | 14.8 [12.7 to 17.1] | 15.0 [10.1 to 21.2] | 15.4 [11.8 to 19.6]
  New/worsened muscle pain | 38.7 [33.6 to 44.1] | 43.5 [38.2 to 48.8] | 43.2 [37.9 to 48.6] | 41.8 [38.8 to 44.9] | 43.9 [36.4 to 51.7] | 40.5 [35.3 to 45.8]
  New/worsened joint pain | 23.4 [19.0 to 28.1] | 27.3 [22.7 to 32.2] | 23.9 [19.5 to 28.8] | 24.9 [22.3 to 27.6] | 24.3 [18.1 to 31.4] | 22.2 [18.0 to 26.9]
  Use of antipyretic/analgesic medication | 41.9 [36.7 to 47.2] | 43.8 [38.5 to 49.1] | 46.4 [41.1 to 51.8] | 44.0 [41.0 to 47.1] | 51.4 [43.7 to 59.1] | 43.6 [38.3 to 49.0]

11. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Dose 3: Booster Study
Description: Systemic events were reported using an electronic diary. Fever was defined as temperature >=38.0 C and categorized as >=38.0 to 38.4 C; >38.4 to 38.9 C; >38.9 to 40.0 C; >40.0 C. Systemic events including fever, fatigue, headache, chills, new or worsened muscle pain, new or worsened joint pain, vomiting, diarrhea, and use of antipyretic/analgesic medication after Dose 3 were reported.
Time Frame: Within 7 days after Dose 3
Population: Safety population included all randomized participants who received dose 3 of the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Number analyzed (Participants) | 31 | 31
Percentage of participants
  Fever >=38.0 C | 3.2 [0.1 to 16.7] | 6.5 [0.8 to 21.4]
  Fever >=38.0 C to 38.4 C | 0 [0.0 to 11.2] | 6.5 [0.8 to 21.4]
  Fever >38.4 C to 38.9 C | 3.2 [0.1 to 16.7] | 0 [0.0 to 11.2]
  Fever >38.9 C to 40.0 C | 0 [0.0 to 11.2] | 0 [0.0 to 11.2]
  Fever >40.0 C | 0 [0.0 to 11.2] | 0 [0.0 to 11.2]
  Fatigue | 67.7 [48.6 to 83.3] | 83.9 [66.3 to 94.5]
  Headache | 41.9 [24.5 to 60.9] | 58.1 [39.1 to 75.5]
  Chills | 25.8 [11.9 to 44.6] | 19.4 [7.5 to 37.5]
  Vomiting | 3.2 [0.1 to 16.7] | 0 [0.0 to 11.2]
  Diarrhea | 16.1 [5.5 to 33.7] | 6.5 [0.8 to 21.4]
  New/worsened muscle pain | 41.9 [24.5 to 60.9] | 19.4 [7.5 to 37.5]
  New/worsened joint pain | 12.9 [3.6 to 29.8] | 12.9 [3.6 to 29.8]
  Use of antipyretic/analgesic medication | 32.3 [16.7 to 51.4] | 35.5 [19.2 to 54.6]

12. Primary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) From Dose 1 to 1 Month After Dose 2: Primary Study
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly or that was considered to be an important medical event.
Time Frame: Day 1 of Dose 1 up to 1 Month after Dose 2 (for a maximum of 2 months)
Population: Safety population included all randomized participants who received at least 1 dose of the study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | BNT162b2 30 mcg: US Lot 1 | BNT162b2 30 mcg: US Lot 2 | BNT162b2 30 mcg: US Lot 3 | Pooled US Lots | BNT162b2 30 mcg: EU Lot | BNT162b2 20 mcg: US Lot 1
Number analyzed (Participants) | 351 | 352 | 346 | 1049 | 173 | 351
Percentage of participants
  AEs | 5.4 | 6.0 | 5.2 | 5.5 | 10.4 | 6.8
  SAEs | 0 | 0 | 0.3 | 0.1 | 0.6 | 0

13. Primary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) From Dose 3 to 1 Month After Dose 3: Booster Study
Description: as for outcome 12
Time Frame: From Dose 3 to 1 Month after Dose 3 (for a maximum of 35 days)
Population: Safety population included all randomized participants who received Dose 3 of the study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Number analyzed (Participants) | 31 | 31
Percentage of participants
  AEs | 6.5 | 3.2
  SAEs | 0 | 0

14. Primary Outcome: Geometric Mean Titers (GMTs) of SARS-CoV-2 Reference-strain at Baseline: Booster Study
Description: GMTs and 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ were set to 0.5 × LLOQ.
Time Frame: Baseline (prior to Dose 1 of Primary study)
Population: Booster evaluable immunogenicity population: Participants who received 2 doses of vaccine in primary study, Dose 2 - primary study, Dose 3 - booster study within predefined window, had at least 1 valid immunogenicity result from blood sample collected within appropriate window at 1 month after Dose 3, were negative for both SARS-CoV-2 test at Dose 1,1-month post Dose 2, 3, and had no other protocol deviations determined by clinician. Here, "N" = participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Number analyzed (Participants) | 27 | 25
Titer | 20.5 [20.5 to 20.5] | 20.5 [20.5 to 20.5]

15. Primary Outcome: Geometric Mean Titers (GMTs) of SARS-CoV-2 Reference-strain 1 Month After Dose 2: Booster Study
Description: as for outcome 14
Time Frame: 1 Month after Dose 2 of primary study
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Number analyzed (Participants) | 27 | 25
Titer | 971.4 [750.5 to 1257.4] | 749.0 [575.2 to 975.3]

16. Primary Outcome: Geometric Mean Titers (GMTs) of SARS-CoV-2 Reference-strain Before Dose 3: Booster Study
Description: as for outcome 14
Time Frame: Before Dose 3
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Number analyzed (Participants) | 27 | 26
Titer | 263.5 [186.9 to 371.3] | 224.2 [176.4 to 285.1]

17. Primary Outcome: Geometric Mean Titers (GMTs) of SARS-CoV-2 Reference-strain 1 Week After Dose 3: Booster Study
Description: as for outcome 14
Time Frame: 1 Week after Dose 3
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Number analyzed (Participants) | 27 | 26
Titer | 2159.3 [1568.4 to 2972.8] | 1283.4 [939.4 to 1753.5]

18. Primary Outcome: Geometric Mean Titers (GMTs) of SARS-CoV-2 Reference-strain 1 Month After Dose 3: Booster Study
Description: as for outcome 14
Time Frame: 1 Month after Dose 3
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Number analyzed (Participants) | 27 | 26
Titer | 2035.5 [1502.2 to 2758.1] | 943.3 [699.1 to 1272.7]

19. Primary Outcome: Geometric Mean Titers (GMTs) of SARS-CoV-2 B.1.351-strain at Baseline: Booster Study
Description: GMTs and 2-sided 95% CIs were planned to be calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution).
Time Frame: Baseline (prior to Dose 1 of Primary study)
Population: Data for this outcome was not analyzed as the immunogenicity samples were not tested for SARS-CoV-2 B.1.351-strain at Baseline as the South African strain was no longer of clinical interest and required responses have been well understood from other studies.
Arm/Group | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Number analyzed (Participants) | 0 | 0

20. Primary Outcome: Geometric Mean Titers (GMTs) of SARS-CoV-2 B.1.351-strain 1 Month After Dose 2: Booster Study
Description: as for outcome 19
Time Frame: 1 Month after Dose 2 of primary study
Population: Data for this outcome was not analyzed as the immunogenicity samples were not tested for SARS-CoV-2 B.1.351-strain at 1 month after dose 2 as the South African strain was no longer of clinical interest and required responses have been well understood from other studies.
Arm/Group | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Number analyzed (Participants) | 0 | 0

21. Primary Outcome: Geometric Mean Titers (GMTs) of SARS-CoV-2 B.1.351-strain Before Dose 3: Booster Study
Description: as for outcome 14
Time Frame: Before Dose 3
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Number analyzed (Participants) | 27 | 26
Titer | 103.0 [75.4 to 140.8] | 94.0 [67.5 to 130.8]

22. Primary Outcome: Geometric Mean Titers (GMTs) of SARS-CoV-2 B.1.351-strain 1 Week After Dose 3: Booster Study
Description: as for outcome 14
Time Frame: 1 Week after Dose 3
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Number analyzed (Participants) | 27 | 26
Titer | 1614.1 [1172.8 to 2221.6] | 1729.8 [1160.0 to 2579.4]

23. Primary Outcome: Geometric Mean Titers (GMTs) of SARS-CoV-2 B.1.351-strain 1 Month After Dose 3: Booster Study
Description: as for outcome 14
Time Frame: 1 Month after Dose 3
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Number analyzed (Participants) | 27 | 26
Titer | 1358.4 [968.5 to 1905.1] | 1411.1 [950.1 to 2095.9]

24. Primary Outcome: Geometric Mean Concentrations (GMCs) of Full-length S-binding IgG Levels at Baseline: Booster Study
Description: GMCs were calculated by exponentiating the mean logarithm of the concentrations and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ were set to 0.5*LLOQ.
Time Frame: Baseline (prior to Dose 1 of Primary study)
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Unit per milliliter
Arm/Group | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Number analyzed (Participants) | 27 | 26
Unit per milliliter | 3.4 [2.0 to 5.7] | 3.4 [2.3 to 5.1]

25. Primary Outcome: Geometric Mean Concentrations (GMCs) of Full-length S-binding IgG Levels 1 Month After Dose 2: Booster Study
Description: as for outcome 24
Time Frame: 1 Month after Dose 2 of primary study
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Unit per milliliter
Arm/Group | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Number analyzed (Participants) | 27 | 26
Unit per milliliter | 6529.1 [5212.9 to 8177.6] | 3796.9 [1899.8 to 7588.4]

26. Primary Outcome: Geometric Mean Concentrations (GMCs) of Full-length S-binding IgG Levels Before Dose 3: Booster Study
Description: as for outcome 24
Time Frame: Before Dose 3
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Unit per milliliter
Arm/Group | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Number analyzed (Participants) | 27 | 26
Unit per milliliter | 1834.5 [1458.5 to 2307.5] | 1851.6 [1441.9 to 2377.8]

27. Primary Outcome: Geometric Mean Concentrations (GMCs) of Full-length S-binding IgG Levels 1 Week After Dose 3: Booster Study
Description: as for outcome 24
Time Frame: 1 Week after Dose 3
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Unit per milliliter
Arm/Group | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Number analyzed (Participants) | 27 | 26
Unit per milliliter | 10756.9 [8478.9 to 13647.0] | 10412.3 [7733.0 to 14020.0]

28. Primary Outcome: Geometric Mean Concentrations (GMCs) of Full-length S-binding IgG Levels 1 Month After Dose 3: Booster Study
Description: as for outcome 24
Time Frame: 1 Month after Dose 3
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Unit per milliliter
Arm/Group | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Number analyzed (Participants) | 27 | 26
Unit per milliliter | 7983.0 [6266.0 to 10170.6] | 6676.9 [5242.6 to 8503.6]

29. Primary Outcome: Geometric Mean Fold Rises (GMFRs) in Full-length S-binding IgG Levels From 1 Month After Dose 2 to 1 Week After Dose 3: Booster Study
Description: GMFRs were defined as ratios of the geometric mean concentration of IgG at 1 week after Dose 3 to the geometric mean concentration of IgG at 1 month after dose 2. GMFRs were calculated by exponentiating the mean logarithm of fold rises and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ were set to 0.5*LLOQ.
Time Frame: From 1 Month after Dose 2 to 1 Week after Dose 3
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Number analyzed (Participants) | 27 | 26
Fold rise | 1.6 [1.3 to 2.0] | 2.7 [1.3 to 5.9]

30. Primary Outcome: Geometric Mean Fold Rises (GMFRs) in Full-length S-binding IgG Levels From 1 Month After Dose 2 to 1 Month After Dose 3: Booster Study
Description: GMFRs were defined as ratios of the geometric mean concentration of IgG at 1 month after Dose 3 to the geometric mean concentration of IgG at 1 month after dose 2. GMFRs were calculated by exponentiating the mean logarithm of fold rises and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ were set to 0.5*LLOQ.
Time Frame: From 1 Month after Dose 2 to 1 Month after Dose 3
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Number analyzed (Participants) | 27 | 26
Fold rise | 1.2 [1.0 to 1.5] | 1.8 [0.9 to 3.6]

31. Primary Outcome: Geometric Mean Fold Rises (GMFRs) in Full-length S-binding IgG Levels Before Dose 3 to 1 Week After Dose 3: Booster Study
Description: GMFRs were defined as ratios of the geometric mean concentration of IgG at 1 week after Dose 3 to the geometric mean concentration of IgG before dose 3. GMFRs were calculated by exponentiating the mean logarithm of fold rises and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ were set to 0.5*LLOQ.
Time Frame: Before Dose 3 to 1 Week after Dose 3
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Number analyzed (Participants) | 27 | 26
Fold rise | 5.9 [4.9 to 7.0] | 5.6 [4.4 to 7.2]

32. Primary Outcome: Geometric Mean Fold Rises (GMFRs) in Full-length S-binding IgG Levels Before Dose 3 to 1 Month After Dose 3: Booster Study
Description: GMFRs were defined as ratios of the geometric mean concentration of IgG at 1 month after Dose 3 to the geometric mean concentration of IgG before dose 3. GMFRs were calculated by exponentiating the mean logarithm of fold rises and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ were set to 0.5*LLOQ.
Time Frame: Before Dose 3 to 1 Month after Dose 3
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Number analyzed (Participants) | 27 | 26
Fold rise | 4.4 [3.7 to 5.2] | 3.6 [2.9 to 4.5]

33. Primary Outcome: Geometric Mean Fold Rise (GMFRs) in SARS-CoV-2 Reference-strain From 1 Month After Dose 2 to 1 Week After Dose 3: Booster Study
Description: GMFRs were defined as ratios of the geometric mean titers of SARS-CoV-2 reference-strain at 1 week after Dose 3 to the geometric mean titers of SARS-CoV-2 reference-strain at 1 month after dose 2. GMFRs were calculated by exponentiating the mean logarithm of fold rises and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ were set to 0.5*LLOQ.
Time Frame: From 1 Month after Dose 2 to 1 Week after Dose 3
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Number analyzed (Participants) | 27 | 25
Fold rise | 2.2 [1.6 to 3.0] | 1.7 [1.3 to 2.2]

34. Primary Outcome: Geometric Mean Fold Rise (GMFRs) in SARS-CoV-2 Reference-strain From 1 Month After Dose 2 to 1 Month After Dose 3: Booster Study
Description: GMFRs were defined as ratios of the geometric mean titers of SARS-CoV-2 reference-strain at 1 month after Dose 3 to the geometric mean titers of SARS-CoV-2 reference-strain at 1 month after dose 2. GMFRs were calculated by exponentiating the mean logarithm of fold rises and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ were set to 0.5*LLOQ.
Time Frame: From 1 Month after Dose 2 to 1 Month after Dose 3
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Number analyzed (Participants) | 27 | 25
Fold rise | 2.1 [1.6 to 2.7] | 1.2 [0.9 to 1.6]

35. Primary Outcome: Geometric Mean Fold Rise (GMFRs) in SARS-CoV-2 Reference-strain Before Dose 3 to 1 Week After Dose 3: Booster Study
Description: GMFRs were defined as ratios of the geometric mean titers of SARS-CoV-2 reference-strain at 1 week after Dose 3 to the geometric mean titers of SARS-CoV-2 reference-strain before dose 3. GMFRs were calculated by exponentiating the mean logarithm of fold rises and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ were set to 0.5*LLOQ.
Time Frame: Before Dose 3 to 1 Week after Dose 3
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Number analyzed (Participants) | 27 | 26
Fold rise | 8.2 [5.3 to 12.7] | 5.7 [4.5 to 7.3]

36. Primary Outcome: Geometric Mean Fold Rise (GMFRs) in SARS-CoV-2 Reference-strain Before Dose 3 to 1 Month After Dose 3: Booster Study
Description: GMFRs were defined as ratios of the geometric mean titers of SARS-CoV-2 reference-strain at 1 month after Dose 3 to the geometric mean titers of SARS-CoV-2 reference-strain before dose 3. GMFRs were calculated by exponentiating the mean logarithm of fold rises and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ were set to 0.5*LLOQ.
Time Frame: Before Dose 3 to 1 Month after Dose 3
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Number analyzed (Participants) | 27 | 26
Fold rise | 7.7 [5.6 to 10.7] | 4.2 [3.2 to 5.5]

37. Primary Outcome: Geometric Mean Fold Rise (GMFRs) in SARS-CoV-2 B.1.351-strain From 1 Month After Dose 2 to 1 Week After Dose 3: Booster Study
Description: GMFRs were defined as ratios of the geometric mean titers of SARS-CoV-2 B.1.351-strain at 1 week after Dose 3 to the geometric mean titers of SARS-CoV-2 B.1.351-strain at 1 month after dose 2. GMFRs were planned to be calculated by exponentiating the mean logarithm of fold rises and the corresponding CIs (based on the Student t distribution).
Time Frame: From 1 Month after Dose 2 to 1 Week after Dose 3
Population: Data for this outcome was not analyzed as the immunogenicity samples from 1 month after dose 2 were not tested for SARS-CoV-2 B.1.351-strain as the South African strain was no longer of clinical interest and required responses have been well understood from other studies.
Arm/Group | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Number analyzed (Participants) | 0 | 0

38. Primary Outcome: Geometric Mean Fold Rise (GMFRs) in SARS-CoV-2 B.1.351-strain From 1 Month After Dose 2 to 1 Month After Dose 3: Booster Study
Description: GMFRs were defined as ratios of the geometric mean titers of SARS-CoV-2 B.1.351-strain at 1 month after Dose 3 to the geometric mean titers of SARS-CoV-2 B.1.351-strain at 1 month after dose 2. GMFRs were planned to be calculated by exponentiating the mean logarithm of fold rises and the corresponding CIs (based on the Student t distribution).
Time Frame: From 1 Month after Dose 2 to 1 Month after Dose 3
Population: as for outcome 20
Arm/Group | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Number analyzed (Participants) | 0 | 0

39. Primary Outcome: Geometric Mean Fold Rise (GMFRs) in SARS-CoV-2 B.1.351-strain Before Dose 3 to 1 Week After Dose 3: Booster Study
Description: GMFRs were defined as ratios of the geometric mean titers of SARS-CoV-2 B.1.351-strain at 1 week after Dose 3 to the geometric mean titers of SARS-CoV-2 B.1.351-strain before dose 3. GMFRs were calculated by exponentiating the mean logarithm of fold rises and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ were set to 0.5*LLOQ.
Time Frame: Before Dose 3 to 1 Week after Dose 3
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Number analyzed (Participants) | 27 | 26
Fold rise | 15.7 [11.2 to 22.0] | 18.4 [13.8 to 24.6]

40. Primary Outcome: Geometric Mean Fold Rise (GMFRs) in SARS-CoV-2 B.1.351-strain Before Dose 3 to 1 Month After Dose 3: Booster Study
Description: GMFRs were defined as ratios of the geometric mean titers of SARS-CoV-2 B.1.351-strain at 1 month after Dose 3 to the geometric mean titers of SARS-CoV-2 B.1.351-strain before dose 3. GMFRs were calculated by exponentiating the mean logarithm of fold rises and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ were set to 0.5*LLOQ.
Time Frame: Before Dose 3 to 1 Month after Dose 3
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Number analyzed (Participants) | 27 | 26
Fold rise | 13.2 [9.6 to 18.1] | 15.0 [11.3 to 19.9]

41. Primary Outcome: Percentage of Participants With Seroresponse to Reference Strain at 1 Month After Dose 2: Booster Study
Description: Seroresponse was defined as greater than equal to (>=) 4-fold increase from baseline (before Dose 1 in primary study) to the specified time point. If the baseline measurement was below LLOQ, a post vaccination measurement of >=4*LLOQ was considered a seroresponse. Exact 2-sided 95% CI was based on the Clopper and Pearson method.
Time Frame: 1 Month after Dose 2
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Number analyzed (Participants) | 27 | 25
Percentage of participants | 100 [87.2 to 100.0] | 100 [86.3 to 100.0]

42. Primary Outcome: Percentage of Participants With Seroresponse to Reference Strain Before Dose 3: Booster Study
Description: Seroresponse was defined as >=4-fold increase from baseline (before Dose 1 in primary study) to the specified time point. If the baseline measurement was below LLOQ, a post vaccination measurement of >=4*LLOQ was considered a seroresponse. Exact 2-sided 95% CI was based on the Clopper and Pearson method.
Time Frame: Before Dose 3
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Number analyzed (Participants) | 27 | 25
Percentage of participants | 92.6 [75.7 to 99.1] | 92.0 [74.0 to 99.0]

43. Primary Outcome: Percentage of Participants With Seroresponse to Reference Strain 1 Week After Dose 3: Booster Study
Description: as for outcome 42
Time Frame: 1 Week after Dose 3
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Number analyzed (Participants) | 27 | 25
Percentage of participants | 100.0 [87.2 to 100.0] | 100.0 [86.3 to 100.0]

44. Primary Outcome: Percentage of Participants With Seroresponse to Reference Strain 1 Month After Dose 3: Booster Study
Description: as for outcome 42
Time Frame: 1 Month after Dose 3
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Number analyzed (Participants) | 27 | 25
Percentage of participants | 100.0 [87.2 to 100.0] | 100.0 [86.3 to 100.0]

45. Primary Outcome: Percentage of Participants With Seroresponse to B.1.351 Variant Strain at 1 Month After Dose 2: Booster Study
Description: Seroresponse was defined as >=4-fold increase from baseline (before Dose 1 in primary study) to the specified time point.
Time Frame: 1 Month after Dose 2
Population: Data for this outcome was not analyzed as the immunogenicity samples were not tested for SARS-CoV-2 B.1.351-strain at baseline and 1 month after dose 2 as the South African strain was no longer of clinical interest and required responses have been well understood from other studies.
Arm/Group | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Number analyzed (Participants) | 0 | 0

46. Primary Outcome: Percentage of Participants With Seroresponse to B.1.351 Variant Strain Before Dose 3: Booster Study
Description: as for outcome 45
Time Frame: Before Dose 3
Population: as for outcome 19
Arm/Group | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Number analyzed (Participants) | 0 | 0

47. Primary Outcome: Percentage of Participants With Seroresponse to B.1.351 Variant Strain 1 Week After Dose 3: Booster Study
Description: as for outcome 45
Time Frame: 1 Week after Dose 3
Population: as for outcome 19
Arm/Group | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Number analyzed (Participants) | 0 | 0

48. Primary Outcome: Percentage of Participants With Seroresponse to B.1.351 Variant Strain 1 Month After Dose 3: Booster Study
Description: as for outcome 45
Time Frame: 1 Month after Dose 3
Population: as for outcome 19
Arm/Group | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
Number analyzed (Participants) | 0 | 0

49. Secondary Outcome: Geometric Mean Concentrations (GMCs) of Full-Length S-Binding IgG Levels at Baseline and 1 Month After Dose 2 for 30 mcg Dose of BNT162b2: Primary Study
Description: GMCs were calculated by exponentiating the mean logarithm of the concentrations and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ were set to 0.5* LLOQ.
Time Frame: Baseline (before Dose 1), 1 Month after Dose 2
Population: Evaluable immunogenicity population: Participants who received 2 doses of vaccine in primary study, with Dose 2 received within predefined window, had at least 1 valid immunogenicity result from blood sample collected within an appropriate window at 1 month after Dose 2, were negative for both SARS-CoV-2 test during study and had no other protocol deviations determined by clinician. Here, N=participants evaluable for this outcome measure and n=participants evaluable at specified time points.
Measure: Geometric Mean (95% Confidence Interval); unit: Unit per milliliter
Arm/Group | BNT162b2 30 mcg: US Lot 1 | BNT162b2 30 mcg: US Lot 2 | BNT162b2 30 mcg: US Lot 3 | Pooled US Lots | BNT162b2 30 mcg: EU Lot
Number analyzed (Participants) | 324 | 311 | 310 | 945 | 160
Unit per milliliter
  Baseline: number analyzed (Participants) | 323 | 311 | 310 | 944 | 160
  Baseline | 3.1 [2.7 to 3.5] | 2.6 [2.3 to 3.0] | 2.6 [2.2 to 3.0] | 2.8 [2.5 to 3.0] | 2.6 [2.1 to 3.2]
  1 Month After Dose 2 | 6269.8 [5717.7 to 6875.2] | 6222.3 [5721.5 to 6766.9] | 6818.9 [6280.9 to 7403.1] | 6428.7 [6116.6 to 6756.8] | 6098.9 [5446.0 to 6830.1]

50. Secondary Outcome: Geometric Mean Fold Rises (GMFRs) in Full-Length S-Binding lgG Levels From Baseline to 1 Month After Dose 2 for 30 mcg Dose of BNT162b2: Primary Study
Description: GMFRs were defined as ratios of the geometric mean concentration of IgG at 1 month after Dose 2 to the geometric mean concentration of IgG at Baseline. GMFRs were calculated by exponentiating the mean logarithm of fold rises and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ were set to 0.5*LLOQ.
Time Frame: From Baseline (before Dose 1) up to 1 Month after Dose 2
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | BNT162b2 30 mcg: US Lot 1 | BNT162b2 30 mcg: US Lot 2 | BNT162b2 30 mcg: US Lot 3 | Pooled US Lots | BNT162b2 30 mcg: EU Lot
Number analyzed (Participants) | 323 | 311 | 310 | 944 | 160
Fold rise | 2036.6 [1744.5 to 2377.7] | 2367.1 [2028.6 to 2762.2] | 2645.2 [2271.2 to 3080.8] | 2331.9 [2133.7 to 2548.5] | 2373.8 [1901.2 to 2963.9]

51. Secondary Outcome: Geometric Mean Titers (GMT) of SARS-CoV-2 Neutralizing Titers at Baseline and 1 Month After Dose 2 for 20 mcg and 30 mcg Dose of BNT162b2 From US Lot 1: Primary Study
Description: GMTs and 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ were set to 0.5* LLOQ.
Time Frame: Baseline (before Dose 1), 1 Month after Dose 2
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | BNT162b2 30 mcg: US Lot 1 | BNT162b2 20 mcg: US Lot 1
Number analyzed (Participants) | 324 | 318
Titer
  Baseline | 20.5 [20.5 to 20.5] | 20.5 [20.5 to 20.5]
  1 Month after Dose 2 | 969.6 [905.7 to 1038.0] | 913.0 [843.4 to 988.3]

52. Secondary Outcome: Geometric Mean Fold Rises (GMFRs) in SARS-CoV-2 Neutralizing Titers From Baseline to 1 Month After Dose 2 for 20 mcg and 30 mcg Dose of BNT162b2 From US Lot 1: Primary Study
Description: GMFRs were defined as ratios of the geometric mean titers of SARS-CoV-2 at 1 month after Dose 2 to the geometric mean titers of SARS-CoV-2 at Baseline. GMFRs were calculated by exponentiating the mean logarithm of fold rises and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ were set to 0.5* LLOQ.
Time Frame: From Baseline (before Dose 1) up to 1 Month after Dose 2
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | BNT162b2 30 mcg: US Lot 1 | BNT162b2 20 mcg: US Lot 1
Number analyzed (Participants) | 324 | 318
Fold rise | 47.3 [44.2 to 50.6] | 44.5 [41.1 to 48.2]

ADVERSE EVENTS:
Time Frame: AEs and SAEs-For primary study: From Dose 1 to 1 Month after Dose 2 (up to a maximum of 2 months); For booster study: From Dose 3 to 1 Month after Dose 3 (up to a maximum of 35 days); Local reactions/systemic events: Within 7 days after each dose
Description: Safety population: participants who received at least 1 dose and had safety data available. AEs included events collected in electronic diary (local and systemic reactions; systematic assessment) and events collected on case report form at each visit (non-systematic assessment). 1 participant randomized to US Lot 1 was administered US Lot 1 for Dose 1 and US Lot 3 for Dose 2, therefore, the participant was included in both reporting groups (US Lot 1 and US Lot 3) for non-SAEs.
Arm/Group | BNT162b2 30 mcg: US Lot 1 | BNT162b2 30 mcg: US Lot 2 | BNT162b2 30 mcg: US Lot 3 | BNT162b2 30 mcg: EU Lot | BNT162b2 20 mcg: US Lot 1 | BNT162b2 30 mcg: Booster Dose | BNT162b2.B.1.351 30 mcg: Booster Dose
All-Cause Mortality (participants affected / at risk) | 0/351 | 0/352 | 0/346 | 0/173 | 0/351 | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/351 | 0/352 | 1/346 | 1/173 | 0/351 | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 341/351 | 336/352 | 335/347 | 165/173 | 342/351 | 30/31 | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BNT162b2 30 mcg: US Lot 1 (N=351) | BNT162b2 30 mcg: US Lot 2 (N=352) | BNT162b2 30 mcg: US Lot 3 (N=346) | BNT162b2 30 mcg: EU Lot (N=173) | BNT162b2 20 mcg: US Lot 1 (N=351) | BNT162b2 30 mcg: Booster Dose (N=31) | BNT162b2.B.1.351 30 mcg: Booster Dose (N=31)
Migrainosus (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BNT162b2 30 mcg: US Lot 1 (N=351) | BNT162b2 30 mcg: US Lot 2 (N=352) | BNT162b2 30 mcg: US Lot 3 (N=347) | BNT162b2 30 mcg: EU Lot (N=173) | BNT162b2 20 mcg: US Lot 1 (N=351) | BNT162b2 30 mcg: Booster Dose (N=31) | BNT162b2.B.1.351 30 mcg: Booster Dose (N=31)
Diarrhoea (Gastrointestinal disorders) | 57 | 50 | 48 | 26 | 54 | 5 | 2
Vomiting (Gastrointestinal disorders) | 10 | 7 | 12 | 4 | 8 | 1 | 0
Chills (General disorders) | 115 | 120 | 129 | 56 | 92 | 8 | 6
Fatigue (General disorders) | 276 | 259 | 281 | 133 | 265 | 21 | 26
Injection site erythema (General disorders) | 16 | 19 | 23 | 8 | 16 | 3 | 1
Injection site pain (General disorders) | 319 | 302 | 316 | 158 | 314 | 28 | 29
Injection site swelling (General disorders) | 21 | 31 | 25 | 8 | 22 | 2 | 2
Pyrexia (General disorders) | 26 | 22 | 29 | 16 | 20 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 82 | 96 | 83 | 42 | 78 | 4 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 136 | 153 | 150 | 76 | 142 | 13 | 6
Headache (Nervous system disorders) | 234 | 229 | 223 | 119 | 224 | 13 | 18
Syncope (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Benign abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 3 | 2 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-05-03): https://cdn.clinicaltrials.gov/large-docs/53/NCT04713553/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/53/NCT04713553/SAP_001.pdf